CLINICAL TRIAL: NCT02075866
Title: Finnish Genetic Study for Arrhythmic Events
Acronym: FinGesture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Other Study IDs: Uoulu-FinGesture
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Sudden Cardiac Death; Acute Coronary Event
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

SUMMARY:
Finnish Genetic Study for Arrhythmic Events (FinGesture is a prospective case-control study assessing the characteristics and genetic background of consecutive series of autopsy verified out-of-hospital victims of SCD vs. survivors of an acute coronary event in a specific geographical area in northern Finland.

ELIGIBILITY:
Inclusion Criteria:

* Sudden cardiac death verified by medicolegal autopsy (cases)
* Acute coronary event (increased troponin levels/ECG markers of ischemia/angina pectoris; two out of three criteria) (controls).

Exclusion Criteria:

* Sudden death due to other causes (cases).
* Acute coronary event patients who died during hospitalization (controls).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive victims of sudden cardiac death verified by medicolegal autopsy (cases).
  Acute coronary event patients admitted to the Oulu University Hospital who survived to be discharged from the hospital (controls).
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 1998-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
sudden cardiac death | 20 years

CONTACTS AND LOCATIONS:
Locations (1):
- Oulu University Hospital, Oulu, Finland